CLINICAL TRIAL: NCT00572767
Title: Evaluation of the Therapeutic Effect of Amphetamine in Association to Physiotherapy on Motor Recovery After Stroke: a Randomised, Double-Blinded, Placebo-Controlled Trial
Brief Title: Evaluation of the Effect of Dextro-Amphetamin Added to Physiotherapy in Patients After Stroke
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Intended length of study ended
Sponsor: Reha Rheinfelden (Other)
Responsible Party: Ettlin, Th. Prof., Reha Rheinfelden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000/001; 2000/030
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Stroke
Keywords: randomised-controlled trial; ischemic stroke; motor recovery; amphetamine; motor recovery of patients after a first-ever ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Dextro-Amphetamin
- 2 (Placebo Comparator)
  Interventions: Other: Glucose

INTERVENTIONS:
Drug: Dextro-Amphetamin — After a two week baseline phase the patients will receive a dose of 10mg Dexamphetamine on two days per week for five weeks. Within a time frame of one to three hours they should receive physiotherapy focusing on neurodevelopmental (NDT) for one hour.
  Arms: 1
Other: Glucose — After a two week baseline phase the patients will receive a dose of 10mg of a placebo (same appearance as the experimental drug) on two days per week for five weeks. Within a time frame of one to three hours they should receive physiotherapy focusing on neurodevelopmental (NDT) for one hour.
  The treatment of the control group will be the same as for the experimental group except the content of the drug capsule.
  Arms: 2

SUMMARY:
The aim of the study is to evaluate the effect of Dextro-amphetamin added to physiotherapy on motor recovery in patients after stroke. The study is a double-blinded placebo-controlled randomised controlled trial.

Patients after a first-ever ischemic stroke will receive Dexamphetamine (10mg) twice per week for a duration of five weeks after a baseline phase of two weeks.

The outcome measure focuses on motor recovery and will be assessed:

* one and two weeks before study intervention (baseline phase)
* five times during the study intervention
* one week after study intervention (follow-up)
* once after six and twelve months after start of the study intervention (follow-up).

ELIGIBILITY:
Inclusion Criteria:

* patients after first-ever ischemic stroke with a clinical relevant paresis of the upper and lower limb (general clinical muscle testing below level four)
* correlation of clinical symptoms with a brain imaging (CT or MRI)
* able to communicate with the neurological examiner and understand the aim/matter of the study (with or without aphasia)
* start of the first oral application of the study drug between the fourteenth and 60th day after stroke onset
* older than 13 years
* given written informed consent (or two independent witnesses)

Exclusion Criteria:

* intracranial or (chronic) subdural hemorrhages
* any additional neurological or psychiatric illnesses
* instable arrythmia
* not controlled or treated arterial hypertension
* ensured cardioembolic event
* anxiolytica, neuroleptica, or alpha-adrenergic antagonists or agonists respectively
* certain anticonvulsiva or antihypertonica
* manifest hyperthyreosis
* dementia or terminal illnesses
* epilepsy, phaeochromocytoma or glaucoma
* women known to be pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2001-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Chedoke-McMaster Stroke Assessment (motor impairment measure) | Over the whole duration of the study (2001 to 2006, ten times for each patient)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry M. Ettlin, Prof., Principal Investigator — Reha Rheinfelden
Locations (1):
- Reha Rheinfelden, Rheinfelden, Canton of Aargau, Switzerland

REFERENCES:
- [Derived] Schuster C, Maunz G, Lutz K, Kischka U, Sturzenegger R, Ettlin T. Dexamphetamine improves upper extremity outcome during rehabilitation after stroke: a pilot randomized controlled trial. Neurorehabil Neural Repair. 2011 Oct;25(8):749-55. doi: 10.1177/1545968311405674. Epub 2011 Jun 28. PMID 21712481